CLINICAL TRIAL: NCT00002592
Title: AUTOLOGOUS BONE MARROW TRANSPLANTATION USING C-MYB (LR-3001) ANTISENSE OLIGODEOXYNUCLEOTIDE TREATED BONE MARROW IN CHRONIC MYELOGENOUS LEUKEMIA IN CHRONIC OR ACCELERATED PHASE
Brief Title: Chemotherapy and Bone Marrow Transplantation in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000063772; UPCC-3492; NCI-H94-0532
Record Dates: First submitted 1999-11-01; First posted 2004-03-26 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Leukemia
Keywords: relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase | interventions — LR 3001; Filgrastim; Busulfan; Cyclophosphamide

INTERVENTIONS:
Biological: c-myb antisense oligonucleotide G4460
Biological: filgrastim
Drug: busulfan
Drug: cyclophosphamide
Procedure: autologous bone marrow transplantation
Procedure: in vitro-treated bone marrow transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with autologous bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy followed by autologous bone marrow transplantation in treating patients with chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the ability of c-myb antisense oligodeoxynucleotide to purge bone marrow cells of clonogenic chronic myelogenous leukemia tumor cells and repopulate the bone marrow with normal stem cells in patients treated with high-dose busulfan and cyclophosphamide followed by autologous bone marrow transplantation using marrow treated with c-myb antisense oligodeoxynucleotide. II. Determine the response rate, degree of hematopoietic reconstitution, overall survival, and relapse-free survival of patients treated with this regimen. III. Determine the toxicity of this regimen in these patients.

OUTLINE: Patients undergo bone marrow harvest. The bone marrow is treated with c-myb antisense oligodeoxynucleotide and cryopreserved. A portion of the marrow is cryopreserved untreated in case of engraftment failure. Patients receive oral busulfan every 6 hours on days -7 to -4 for a total of 16 doses. Patients receive cyclophosphamide IV over 1 hour on days -3 and -2. Bone marrow is reinfused on day 0. Patients receive filgrastim (G-CSF) subcutaneously daily beginning on day 0 and continuing until blood counts recover. Patients are followed every 2-3 months for 2 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically and cytologically proven chronic myelogenous leukemia Accelerated phase OR Chronic phase No hypocellular marrow (less than 25% cellularity) No patients under age 55 with a HLA-matched sibling donor

PATIENT CHARACTERISTICS: Age: 18 to 60 Performance status: 0-1 Hematopoietic: Granulocyte count greater than 1,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL AST less than 3 times normal Renal: Creatinine less than 2.0 mg/dL Creatinine clearance greater than 60 mL/min Cardiovascular: Left ventricular ejection fraction normal No significant cardiac disease requiring digoxin, diuretics, antiarrhythmics, or antianginal medications Pulmonary: PFTs normal DLCO normal Other: No persistent infection requiring antibiotics No concurrent organ damage or medical problem that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 months since prior interferon therapy Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 1993-06; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Number of Adberse Events

CONTACTS AND LOCATIONS:
Overall Officials: Selina M. Luger, MD, Study Chair — Abramson Cancer Center at Penn Medicine
Locations (1):
- University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania, United States